CLINICAL TRIAL: NCT03598140
Title: Sildenafil Treatment for Traumatic Vascular Injury in Athletes
Brief Title: Sildenafil Treatment for Mild TBI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI, Dr. Josh Gaston, left the institution and the study has been stopped.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kan Ding, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 032018-063
Record Dates: First submitted 2018-06-11; First posted 2018-07-26 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Vascular System Injuries; Concussion, Brain; Post-Concussion Syndrome
Keywords: Sildenafil; Concussion; CBF; CVR
MeSH Terms: conditions — Vascular System Injuries; Brain Concussion; Post-Concussion Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: This study is a placebo-controlled, double-blinded clinical trial. Randomization will be 1:1 sildenafil:placebo, and will be in blocks of 10. In this study, 100 boxers and 80 controls will be enrolled and randomized.
Who Masked: Participant, Investigator
Masking Description: Investigators associated with this study will not have access to the randomization schedule. The principal investigator, study team, and study subjects will be blinded in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo oral capsule (Placebo Comparator): If randomized to placebo, the participant will receive single (Group 1) or multiple (once-a-day for 14 days; Group 2) treatments.
  Interventions: Drug: Placebo oral capsule
- Sildenafil Citrate (Active Comparator): If randomized to sildenafil (60mg), the participant will receive single (Group 1) or multiple (once-a-day for 14 days; Group 2) treatments.
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate — Sildenafil 60mg once (Group 1) or daily for 2 weeks (Group 2)
  Other Names: Viagra
  Arms: Sildenafil Citrate
Drug: Placebo oral capsule — Placebo once (Group 1) or daily for 2 weeks (Group 2)
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
About 300,000 people are hospitalized for traumatic brain injury (TBI) each year. After TBI, secondary brain injury escalates due in part to heightened levels of oxidant injury, inflammation, and vascular injury. Traumatic cerebral vascular injury (TCVI) may begin almost immediately after the primary injury and evolve into chronic neurodegenerative conditions. TCVI is a very complex TBI endophenotype and microvascular injuries have been described in a plethora of animal and human TBI studies. These injuries consist of endothelial injury, disruption of the blood brain barrier (BBB), a reduction of capillary density, intravascular microthrombi, and white-matter degeneration. Recently, use of magnetic resonance imaging (MRI)-Blood Oxygen Level Dependent (BOLD) combined with hypercapnia (high spatial and temporal resolution) by our research group has proven to be more sensitive at measuring alterations of cerebral blood flow (CBF) in TBI subjects. The goal of the proposed research is to test the efficacy of Viagra® (sildenafil) at normalizing CBF and improving cognitive outcomes in people that have experienced a TBI. Sildenafil is a phosphodiesterase-5 (PDE-5) inhibitor that has previously been administered as a therapy for high blood pressure and erectile dysfunction. In people that have been affected by stroke-induce neurotrauma, sildenafil improved CBF and was found to be neuroprotective. With respect to chronic TBI, previous studies have demonstrated that sildenafil therapy potentiates cardiovascular reactivity (CVR) in areas of the brain with damaged endothelium. In this proposal, the investigators will test the hypothesis that sildenafil treatment in boxers/Mixed Martial Arts (MMA) fighters soon after concussion normalizes CBF, potentiates CVR, reduces post-concussion symptoms, and improves cognition.

DETAILED DESCRIPTION:
In this study, 100 professional boxers that experience a concussion will be enrolled, randomized to either placebo or sildenafil (60mg) drug treatment, and arterial spin labeling and BOLD-MRI with hypercapnia will used to assess CBF and CVR, respectively. Symptom reporting, blood biomarkers, and neuropsychological testing will also be conducted. The timepoints for this study are baseline (pre-fight), and once between days 1 and 3 and day 30 after injury.

ELIGIBILITY:
Inclusion Criteria:

For Athletes

1. Age 18-35
2. Male or female professional boxers/MMA fighters
3. Ability to undergo MR imaging procedures
4. At least one of the following:

   1. Knockout (KO)/Technical Knockout (TKO) scored by fight referee.
   2. Greater than 25 blows to the head.
5. Significant post-concussive symptoms (Symptom Score > 1 on at least 3 items from the Rivermead Post-Concussion Questionnaire)

For Controls

1. Age 18-35
2. Male of female who do not participate in contact sports
3. Screen negative for mild TBI (mTBI) using Ohio State TBI Identification

Exclusion Criteria:

1. Contraindication to sildenafil which includes the following:

   1. Current use of organic nitrate vasodilators
   2. Use of ritonavir (HIV-protease inhibitor)
   3. Current use of erythromycin, ketoconazole, or itraconazole
   4. Current use of cimetidine
   5. Current resting hypotension (BP < 90/50 mm Hg)
   6. Current severe renal insufficiency (Creatinine Clearance < 30 milliliters/minute)
   7. Current hepatic cirrhosis
   8. Current cardiac failure or coronary artery disease causing unstable angina
   9. Retinitis pigmentosa
   10. Known hypersensitivity or allergy to sildenafil of any of its components
2. Daily therapy with a PDE5 inhibitor within the past 2 months
3. Immediate hospitalization for severe concussion
4. History of neurological or psychiatric disorder not related to TBI
5. Known inclusion in another interventional clinical trial
6. Subjects with metal implants that would interfere with the MR imaging procedures
7. Sickle cell disease
8. History of priapism

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate
Started | 10 | 11
Completed | 9 | 11
Not Completed | 1 | 0
Not completed — enrolled but didn't start | 1 | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution, all efforts to locate the data have been exhausted and therefore no results are available to be reported
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Arterial Spin Labeling
Description: Prior to and after sildenafil treatment (60mg) cerebral blood flow will be measured in the athletes and healthy controls.
Time Frame: 3 years
Population: as for baseline characteristics
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rivermead Post Concussion Symptoms Questionnaire (RPQ)
Description: This test will measure a range of injury severities:
  0= Not experienced at all
  1. No more of a problem
  2. A mild problem
  3. A moderate problem
  4. A severe problem Improvement or worsening of symptoms (headaches, nausea, fatigue, feeling depressed, light sensitivity, double vision, etc.) will be recorded. The combined score from all symptoms will be recorded at the indicated time-points.
Time Frame: 3 years
Population: as for baseline characteristics
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Hopkins Verbal Learning Task (HVLT)
Description: Using the HVLT, performance in learning and memory will be measured in concussed athletes and healthy controls.
Time Frame: 3 years
Population: as for baseline characteristics
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: BOLD MRI With Hypercapnia
Description: Before and after sildenafil treatment, cerebrovascular reactivity will be measured in the athletes and healthy controls.
Time Frame: 3 years
Population: as for baseline characteristics
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The PI has left the institution, all efforts to locate the data have been exhausted and therefore no adverse events available to be reported
Description: Study closed, all efforts to obtain data have been exhausted, data cannot be reported
Arm/Group | Placebo Oral Capsule | Sildenafil Citrate
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Dr. Gaston who was the initial PI, left the institution and the study has been stopped.The Department was able to manage to report the results that they could gather as the previous PI didn't disclose the information before leaving the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03598140/Prot_SAP_000.pdf